CLINICAL TRIAL: NCT04840693
Title: Genomic and Metabolomic Markers Reflecting the Complications of Hypercortisolism
Brief Title: Genomic and Metabolomic Markers Reflecting the Complications of Hypercortisolism (CUSHINGOMICS)
Acronym: CUSHINGOMICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: European Union's Horizon 2020 research and innovation programme under grant agreement No 633983 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190799; 2020-A02714-35 (Other: ID-RCB)
Record Dates: First submitted 2021-01-12; First posted 2021-04-12 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Adult Glucocorticoid Excess; Adult Adrenal Insufficiency
Keywords: Hypercortisalism; Glucocorticoids excess; Cushing's syndrome
MeSH Terms: conditions — Adrenal Insufficiency; Cushing Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Excess of endogenous glucoglucocorticoids (group 1) (Experimental): v
  Interventions: Biological: Biological samples; Other: Complications
- Exogenous hypercortisolisms (group 2) (Experimental): a disease justifying the up-coming start of a glucocorticoid therapy
  Interventions: Biological: Biological samples; Other: Complications
- Adrenal insufficiency (group 3) (Experimental): chronic adrenal insufficiency
  Interventions: Biological: Biological samples; Other: Complications
- Control (group 4) (Other): without glucocorticoid excess
  Interventions: Biological: Biological samples; Other: Complications

INTERVENTIONS:
Biological: Biological samples — blood, urine, saliva
Other: Complications — bone mineral density, diabetes, hypertension, quality of life (quality of life questionnaire SF-36)

SUMMARY:
The excess of glucocorticoid, whether endogenous or exogenous, results in Cushing's syndrome, associating a particular distribution of fats (accumulation in the face and trunk), a decrease in the thickness of the muscles, diabetes, hypertension or osteoporosis.

The level of effects obviously depends on the extent of the excess glucocorticoids, and on the duration of this exposure. However, the manifestations of Cushing's syndrome also depend very much on the sensitivity of each individual to glucocorticoids for each of these conditions. Indeed, for the same duration and level of exposure, some will have diabetes only, others only osteoporosis, others hypertension, while still others will have these three complications. Today the investigators are unable to specify individual risks. For example, will someone develop diabetes when exposed to glucocorticoids? Or on the contrary will blood sugar level remain normal? The same question arises for hypertension and osteoporosis.

The deficiency of glucocorticoid, called adrenal insufficiency, causes fatigue and discomfort. The intensity of the signs depends on the depth of the insufficiency. Here again, there is a large variability in the sensitivity of each individual to glucocorticoids: when one substitutes for adrenal insufficiency at a given dose, some individuals will feel well, while others will still remain tired. The investigators are unable to specify participant's individual requirement.

The aim of this research is to identify factors that determine individual sensitivity to glucocorticoids. For excess glucocorticoids, the investigators are looking for specific molecular markers for each type of glucocorticoid complication: markers for corticosteroid-induced diabetes, corticosteroid-induced hypertension, or corticosteroid-induced osteoporosis.

For adrenal insufficiency, they are also looking for substitute good balance markers for adrenal insufficiency.

To answer the research question, it is planned to include 400 subjects exposed to glucocorticoid excess (by excess of endogenous glucocorticoids or induced by corticosteroid therapy) and 100 subjects with adrenal insufficiency. It is also planned to include 100 subjects without excess glucocorticoids but presenting either diabetes, hypertension or osteoporosis; these subjects will constitute a control group. The investigators will perform a very large number of measurements in small amounts of blood and urine, in order to identify a few marks specifically associated with each of the complications. This research will identify, for every person exposed to glucocorticoids, the probability of developping some complications, and reversely the probability of being exempt from other complications.

DETAILED DESCRIPTION:
For each participant, easily accessible biological samples will be taken (blood, urine, saliva). From these samples, a large number of molecular markers will be generated (genomics, metabolomics), in search of signatures specifically associated with each complication.

Three main types of complications will be analyzed: diabetes, hypertension and osteoporosis.

The analysis is planned in 4 stages:

* Identify markers for each type of complication in the context of excess frank glucocorticoids, by comparing affected patients and those not affected for each type of complication.
* Subtraction of non-specific markers of diabetes, hypertension and osteoporosis, identified by the analysis of diabetic, hypertensive and osteoporotic patients who do not have excess glucocorticoids
* Test the performance of these markers in an independent cohort of patients presenting an excess of glucocorticoids at variable levels: frank and at least (endogenous, exogenous)
* Test the performance of these markers in a cohort of patients with substituted adrenal insufficiency

ELIGIBILITY:
Inclusion Criteria:

* an endogenous hypercortisolism (group 1)
* a disease justifying the next start of glucocorticoid therapy (group 2)
* chronic adrenal insufficiency (group 3)
* subjects with either diabetes, hypertension or osteoporosis, but without glucocorticoid excess (control group)
* patients will have to be affiliated to a social security scheme
* patients should be able to understand the study and able to express their consent

Exclusion Criteria:

* patients with reduced life expectancy, less than 2 years
* pregnant or lactating women
* patients refusing the protocol
* patients under state medical assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Identification of molecular markers of glucocorticoid-induced hypertension (diagnosed by oscillometric blood pressure), using genomic and metabolomics measurements | 3 years
  Genomic measurements will include whole blood methylome, transcriptome and miRNome. Metabolomic measurements will be performed by mass spectrometry in blood plasma and urine, to characterize a large panel of biochemical compounds. Relevant markers identified with these high throughput methods will be combined into a single multidimensional composite predictor.
Identification of markers of glucocorticoid-induced diabetes (diagnosed by HbA1c), using genomic and metabolomics measurements | 3 years
  Genomic measurements will include whole blood methylome, transcriptome and miRNome. Metabolomic measurements will be performed by mass spectrometry in blood plasma and urine, to characterize a large panel of biochemical compounds. Relevant markers identified with these high throughput methods will be combined into a single multidimensional composite predictor.
Identification of markers of glucocorticoid-induced osteoporosis (diagnosed by bone density test), using genomic and metabolomics measurements | 3 years
  Genomic measurements will include whole blood methylome, transcriptome and miRNome. Metabolomic measurements will be performed by mass spectrometry in blood plasma and urine, to characterize a large panel of biochemical compounds. Relevant markers identified with these high throughput methods will be combined into a single multidimensional composite predictor.

SECONDARY OUTCOMES:
Identification of markers of glucocorticoid-induced depression (diagnosed by a psychiatrist evaluation during routine management), using genomic and metabolomics measurements | 3 years
  Genomic measurements will include whole blood methylome, transcriptome and miRNome. Metabolomic measurements will be performed by mass spectrometry in blood plasma and urine, to characterize a large panel of biochemical compounds. Relevant markers identified with these high throughput methods will be combined into a single multidimensional composite predictor.
Identification of markers of glucocorticoid-induced hypercatabolism (diagnosed clinically: bruising, stretch marks and amyotrophy), using genomic and metabolomics measurements | 3 years
  Genomic measurements will include whole blood methylome, transcriptome and miRNome. Metabolomic measurements will be performed by mass spectrometry in blood plasma and urine, to characterize a large panel of biochemical compounds. Relevant markers identified with these high throughput methods will be combined into a single multidimensional composite predictor.
Identification of markers of glucocorticoid-induced abnormal fat distribution (diagnosed clinically), using genomic and metabolomics measurements | 3 years
  Genomic measurements will include whole blood methylome, transcriptome and miRNome. Metabolomic measurements will be performed by mass spectrometry in blood plasma and urine, to characterize a large panel of biochemical compounds. Relevant markers identified with these high throughput methods will be combined into a single multidimensional composite predictor.
Identification of markers of glucocorticoid-induced thromboembolic episode (diagnosed during routine management), using genomic and metabolomics measurements | 3 years
  Genomic measurements will include whole blood methylome, transcriptome and miRNome. Metabolomic measurements will be performed by mass spectrometry in blood plasma and urine, to characterize a large panel of biochemical compounds. Relevant markers identified with these high throughput methods will be combined into a single multidimensional composite predictor.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newell-Price J, Bertagna X, Grossman AB, Nieman LK. Cushing's syndrome. Lancet. 2006 May 13;367(9522):1605-17. doi: 10.1016/S0140-6736(06)68699-6. PMID 16698415
- [Background] Charmandari E, Nicolaides NC, Chrousos GP. Adrenal insufficiency. Lancet. 2014 Jun 21;383(9935):2152-67. doi: 10.1016/S0140-6736(13)61684-0. Epub 2014 Feb 4. PMID 24503135
- [Background] Overman RA, Yeh JY, Deal CL. Prevalence of oral glucocorticoid usage in the United States: a general population perspective. Arthritis Care Res (Hoboken). 2013 Feb;65(2):294-8. doi: 10.1002/acr.21796. PMID 22807233
- [Background] Fardet L, Petersen I, Nazareth I. Risk of cardiovascular events in people prescribed glucocorticoids with iatrogenic Cushing's syndrome: cohort study. BMJ. 2012 Jul 30;345:e4928. doi: 10.1136/bmj.e4928. PMID 22846415
- [Background] Tauchmanova L, Rossi R, Biondi B, Pulcrano M, Nuzzo V, Palmieri EA, Fazio S, Lombardi G. Patients with subclinical Cushing's syndrome due to adrenal adenoma have increased cardiovascular risk. J Clin Endocrinol Metab. 2002 Nov;87(11):4872-8. doi: 10.1210/jc.2001-011766. PMID 12414841
- See also: Related Info — http://www.ensat-ht.eu/